CLINICAL TRIAL: NCT00210444
Title: A Phase II, Multicentre, Open, Randomised, Parallel Group, Dose Ranging Study to Define the Efficacy of Dysport® in the Treatment of Anal Fissure.
Brief Title: Efficacy Study of Dysport® in the Treatment of Anal Fissure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-38-52120-714
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Anal Fissure
MeSH Terms: conditions — Fissure in Ano | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
To evaluate the effect on healing rates of two different prognostic factors in patients treated with Dysport® for anal fissure: duration of fissure and dose of study drug

ELIGIBILITY:
Inclusion Criteria:

* Patients having idiopathic anal fissure in the posterior anal midline
* Patients having anal fissure present for less than 6 months
* Patients having symptoms (pain) present for a minimum of 2 weeks and not responding after 2 weeks of standard therapy (diet, laxatives, sitz-bathes)

Exclusion Criteria:

* Patients having anal fistulas or anal fissure of various causes such as Crohn disease, Behcet infectious ulceration, anal suppuration, subfissural infiltration, abscesses, acute haemorrhoidal attacks or inflammatory bowel disease
* Patients having idiopathic anal fissure in the anterior anal midline
* Patients having lateral or multiple fissures
* Patients having anal or perianal cancer
* Patients who underwent previous anal surgery or have cicatricial alterations or post-surgical cicatricial lesions
* Patients receiving drugs affecting neuromuscular transmission
* Patients who have received topical anaesthetic within 3 days of injection
* Patients receiving local treatment by myorelaxing agent
* Patients receiving prohibited analgesics
* Patients having bleeding disturbances or currently using coumarin derivates
* Patients having myasthenia or any genetic muscle disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2003-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Healing of the anal fissure by complete re-epithelisation of the anal canal mucosa.

SECONDARY OUTCOMES:
Improvement of anal pain measured by the patients on Analogue Visual Pain Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- Czechia (3):
  - Faculty Nemocnice-III, Brno
  - Faculty Nemocnice, Hradec Králové
  - Thomayer's Memorial Hospital, Prague
- Poland (2):
  - Consulting Room of Proctology, Gdansk
  - Medical University of Lodz, Lodz
- Institute Clinique Fundeni, Bucharest, Romania
- CHU Hopital Charles Nicolle de Tunis, Tunis, Tunisia